CLINICAL TRIAL: NCT02001051
Title: Randomized Control Trial of Adrenalectomy Versus Observation for Subclinical Hypercortisolism
Brief Title: Study of Adrenalectomy Versus Observation for Subclinical Hypercortisolism
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed due to low accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Clinical Center Office of the Associates Director for Radiologic&Imaging Sciences (Unknown)
Responsible Party: Principal Investigator, Dhaval Patel, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140021; 14-C-0021
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-05

CONDITIONS: Subclinical Hypercortisolism; Cushing Syndrome; Adrenal Neoplasm
Keywords: Diabetes, Hypertension, Hypercholesterolemia, Obesity, and Osteoporosis.; Nonoperative and Operative Management; Adrenal Incidentalomas; Excess of Cortisol
MeSH Terms: conditions — Cushing Syndrome; Adrenal Gland Neoplasms; Diabetes Mellitus; Hypertension; Hypercholesterolemia; Obesity; Osteoporosis; Adrenal incidentaloma | interventions — Adrenalectomy; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operative Arm (Other): operative arm
  Interventions: Procedure: Adrenalectomy
- Delayed Operative Arm (Other): delayed operative arm
  Interventions: Other: Observation

INTERVENTIONS:
Procedure: Adrenalectomy — Surgery to remove tumor when enrolled in the protocol.
  Arms: Operative Arm
Other: Observation — Observation for 6 months prior to surgery
  Arms: Delayed Operative Arm

SUMMARY:
Background:

- Adrenal tumors are a common kind of tumor. Some of these secrete extra cortisol into the body, which can lead to diabetes, obesity, and other diseases. Some people with extra cortisol will show symptoms like bruising and muscle weakness. Others will show no signs. This is called subclinical hypercortisolism. Some of these adrenal tumors become malignant. Researchers want to know the best way to treat people with subclinical hypercortisolism. They want to know if removing the tumor by surgery reduces the long-term effects of the disease.

Objectives:

- To see if removing an adrenal tumor by surgery improves blood pressure, diabetes, obesity, osteoporosis, or cholesterol, and cancer detection.

Eligibility:

- Adults 18 and older with an adrenal tumor and high cortisol levels.

Design:

* Participants will be screened with medical history, blood tests, and a computed tomography (CT) scan.
* Participants will have a baseline visit. They will have blood and urine tests and 7 scans. For most scans, a substance is injected through a tube in the arm. Participants will lie still on a table in a machine that takes images.
* Participants will have surgery to remove their tumor. Some will have surgery right away. Some will have surgery 6 months later, after 2 follow-up appointments.
* Participants will have 4 follow-up visits in the first year after surgery. They will have 2 visits the second year, then yearly visits for 3 years. At each follow-up visit, they will have scans and blood tests.

DETAILED DESCRIPTION:
Background:

* Adrenal incidentalomas are common and found in approximately 4-7% of the population.
* About 0.6 to 25% of patients with an adrenal incidentaloma are found to have subclinical hypercortisolism: 2.3% develop subclinical hypercortisolism during follow up and 0.6% develop clinical hypercortisolism during follow up.
* Subclinical hypercortisolism is defined as biochemical excess of cortisol without signs and symptoms of overt hypercortisolism but may be associated with metabolic complications or disease progression and malignancy.
* Overt signs and symptoms of hypercortisolism include facial plethora, easy bruising, violaceous striae, and proximal muscle weakness.
* Several studies suggest that subclinical hypercortisolism may lead to long term consequences such as diabetes, hypertension, hypercholesterolemia, obesity, and osteoporosis.
* Thus, patients with subclinical hypercortisolism may benefit from operative intervention to halt or reverse metabolic complications associated with the disease and the risk of malignant progression.
* The optimal management of patients with subclinical hypercortisolism and adrenal incidentalomas is controversial and no large randomized trial has been conducted.
* We hypothesize that operative treatment would reduce the risk of long term complications of subclinical hypercortisolism and malignant progression, and propose a prospective randomized trial comparing nonoperative and operative management of subclinical hypercortisolism in patients with an adrenal neoplasm.

Objectives:

Primary Endpoints:

-To determine whether unilateral adrenalectomy in patients diagnosed with subclinical hypercortisolism and adrenal neoplasm results in normalization and/or improvement of hypertension as assessed by reduction in pharmacotherapy and/or normalization of blood pressure (systolic pressure <=140 and diastolic pressure <=90), diabetes as assessed by reduction or elimination of pharmacotherapy and/or improvement in A1C to <6.5%, osteoporosis by increase in bone formation markers indicative of increased bone formation, hypercholesterolemia as assessed by a reduction or elimination of pharmacotherapy and/or reduction in low density lipoprotein (LDL) levels to risk-stratified goal levels as defined by Adult Treatment Panel III (ATP III), and/or overweight or obesity as assessed by a 10 percent reduction in weight at 6 months.

Eligibility:

* An individual with an adrenal neoplasm less than 5 cm in size with biochemically confirmed evidence of hypercortisolism (2 out of 3: dexamethasone suppression test (DST) >3 mcgl/dL, elevated urine free cortisol, and/or morning adrenocorticotrophic hormone (ACTH) <2.2 pmol/l) without overt clinical signs and symptoms.
* Age greater than or equal to 18 years.
* Adults must be able to understand and sign the informed consent document.
* Patients must have laboratory and physical examination parameters within acceptable limits based on standard clinical practice.

Design:

* Prospective randomized study comparing adrenalectomy versus observation.
* Patients assigned to the operative arm will undergo adrenalectomy and then followed postoperatively for normalization and/or improvement of metabolic complications associated with hypercortisolism and histologic examination of the resected tumor.
* Patients assigned to the non-operative arm will be monitored for possible complications associated with hypercortisolism for six months, at which point they will cross-over to the operative intervention arm.
* Patients with bilateral adrenal neoplasms will have the larger adrenal neoplasm used as the primary lesion responsible for subclinical hypercortisolism.
* Demographic, clinical, laboratory and pathologic data will be collected for each patient participant. Data will be securely stored in a computerized database.
* Patients will have biochemical testing to determine if their adrenal neoplasm is functioning or nonfunctioning.
* Projected accrual will be 15 to 20 patients per year for a total of 5 years. Thus, we anticipate accruing 62 patients on this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:
* An individual with an adrenal neoplasm less than 5 cm in size with biochemically confirmed evidence of hypercortisolism (2 out of 3: dexamethasone suppression test (DST) >3 mcgl/dL, elevated urine free cortisol, and/or morning adrenocorticotropic hormone (ACTH) <2.2 pmol/l) without overt clinical signs and symptoms.
* Age greater than or equal to 18 years.
* Adults must be able to understand and sign the informed consent document.
* Patients must have laboratory and physical examination parameters within acceptable limits by standard of practice.

EXCLUSION CRITERIA:

* Biochemically and/or radiologically confirmed pheochromocytoma, hyperaldosteronism, or adrenocortical carcinoma.
* Nonfunctioning adrenal neoplasm.
* Pre-existing cancers and/or metastatic disease to the adrenal glands.
* Pregnancy and/or lactation.
* Lack of metabolic complications.
* Imaging features worrisome for malignancy (heterogeneous tumor, presence of calcifications, necrosis, >10 Hounsfield units on an unenhanced computed tomography (CT) scan, and delayed washout of contrast).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-11-27 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2018-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dhaval T Patel, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Toniato A, Merante-Boschin I, Opocher G, Pelizzo MR, Schiavi F, Ballotta E. Surgical versus conservative management for subclinical Cushing syndrome in adrenal incidentalomas: a prospective randomized study. Ann Surg. 2009 Mar;249(3):388-91. doi: 10.1097/SLA.0b013e31819a47d2. PMID 19247023
- [Background] Reincke M. Subclinical Cushing's syndrome. Endocrinol Metab Clin North Am. 2000 Mar;29(1):43-56. doi: 10.1016/s0889-8529(05)70115-8. PMID 10732263
- [Background] Chiodini I. Clinical review: Diagnosis and treatment of subclinical hypercortisolism. J Clin Endocrinol Metab. 2011 May;96(5):1223-36. doi: 10.1210/jc.2010-2722. Epub 2011 Mar 2. PMID 21367932
- [Derived] Neychev V, Steinberg SM, Yang L, Mehta A, Nilubol N, Keil MF, Nieman L, Stratakis CA, Kebebew E. Long-Term Outcome of Bilateral Laparoscopic Adrenalectomy Measured by Disease-Specific Questionnaire in a Unique Group of Patients with Cushing's Syndrome. Ann Surg Oncol. 2015 Dec;22 Suppl 3(Suppl 3):S699-706. doi: 10.1245/s10434-015-4605-1. Epub 2015 May 13. PMID 25968622
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0021.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was enrolled to the delayed operative arm but did not complete. The participant did not have biochemical evidence of subclinical Cushing's and therefore was not eligible.
Groups:
- Delayed Operative Arm Followed by Surgery: delayed operative arm
  Observation: Observation for 6 months prior to surgery
Period: Overall Study
Arm/Group | Operative Arm | Delayed Operative Arm Followed by Surgery
Started | 2 | 2
Completed | 2 | 1
Not Completed | 0 | 1
Not completed — Deemed not eligible following enrollment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Operative Arm | Delayed Operative Arm Followed by Surgery | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.56 (11.68) | 43.25 (12.09) | 45.91 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients That Have Normalization and/or Improvement of Metabolic Complications After Adrenalectomy
Description: Normalization and/or improvement of metabolic complications including hypertension, diabetes, osteoporosis, hypercholesterolemia and/or obesity after adrenalectomy is defined as 35% of patients who improve with surgery versus 5% who do not have surgery.
Time Frame: Assessed at 6 months
Measure: Number; unit: proportion of participants
Arm/Group | Operative Arm | Delayed Operative Arm
Number analyzed (Participants) | 2 | 1
proportion of participants | 1 | 0

2. Primary Outcome: Count of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 39 months and 27 days
Population: No toxicities were experienced by any participants on this trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Operative Arm | Delayed Operative Arm
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

3. Secondary Outcome: Proportion of Patients Who Are Found to Have Adrenal Cancer After Adrenalectomy
Description: Patients who were tested for and found to have adrenal cancer after adrenalectomy.
Time Frame: Assessed at 6 months
Measure: Number; unit: proportion of participants
Arm/Group | Operative Arm | Delayed Operative Arm
Number analyzed (Participants) | 2 | 1
proportion of participants | 0 | 0

4. Secondary Outcome: Proportion of Patients Who Were Diagnosed With Subclinical Hypercortisolism by Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET)/Computed Tomography (CT) Scan
Description: Proportion of patients who were diagnosed with subclinical hypercortisolism by FDG/PET/CT scan.
Time Frame: Assessed at 6 months
Measure: Number; unit: proportion of participants
Arm/Group | Operative Arm | Delayed Operative Arm
Number analyzed (Participants) | 2 | 1
proportion of participants | 1 | 1

5. Secondary Outcome: To Determine the Optimal Diagnostic Test for Subclinical Hypercortisolism
Description: An assessment of whether 1 mg dexamethasone suppression test, basal adrenocorticotropic hormone (ACTH), midnight salivary cortisol, or urinary free cortisol is the optimal test to diagnose patients with subclinical hypercortisolism.
Time Frame: Assessed at 6 months
Population: This outcome measure was not done. Data was collected and not analyzed because we were not able to determine the optimal test since we only had four patients enrolled, and three patients on study (e.g. low accrual). Therefore, we couldn't do a head to head comparison calculating the sensitivity and specificity.
Arm/Group | Operative Arm | Delayed Operative Arm
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Proportion of Patients That Have Improvement in Quality of Life (QOL) After Adrenalectomy Compared to Medical Therapy
Description: QOL questionnaires were provided to participants to assess well being pre and post operatively. Participants take a self-administered questionnaire to assess physical and mental health according to Cushing's Quality of Life Questionnaire. The score has a minimum of 12 and maximum of 60. A higher score indicates an improved quality of life.
Time Frame: Assessed at 6 months
Measure: Number; unit: proportion of participants
Arm/Group | Operative Arm | Delayed Operative Arm
Number analyzed (Participants) | 2 | 1
proportion of participants | 2 | 0

7. Secondary Outcome: Proportion of Patients That Developed Deep Venous Thrombosis With Subclinical Hypercortisolism
Description: Proportion of patients that developed deep venous thrombosis with subclinical hypercortisolism regardless of whether the participants received adrenalectomy or not.
Time Frame: Assessed at 6 months
Measure: Number; unit: proportion of participants
Arm/Group | Operative Arm | Delayed Operative Arm
Number analyzed (Participants) | 2 | 1
proportion of participants | 0 | 0

8. Secondary Outcome: Correlation Between Dermal Thickness and Patients With Subclinical Hypercortisolism
Description: A skin biopsy and skin ultrasound were done to measure the dermal layer of skin to look for a decrease in the thickness of skin as compared to normal values reported in the literature as measured in millimeters of thickness. Diagnostic sensitivity and changes in skin thickness were assessed.
Time Frame: Assessed at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Operative Arm | Delayed Operative Arm
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 39 months and 27 days.
Description: No toxicities were experienced by any participants on this trial.
Arm/Group | Operative Arm | Delayed Operative Arm
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-01-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT02001051/Prot_SAP_ICF_000.pdf